CLINICAL TRIAL: NCT05408832
Title: Re-engineering Precision Therapeutics Through N-of-1 Trials: Personalized Trials for Stress Management Against Standard of Care
Brief Title: Personalized Trials for Stress Management Against Standard of Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Library of Medicine (NLM) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-0968; R01LM012836 (NIH)
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Stress
Keywords: Stress; Personalized; N-of-1; Virtual; Feasibility; Yoga; Walking; Mindfulness

STUDY DESIGN:
Intervention Model Description: Mixed between and within (Crossover) participant assignment. The study uses a between participant randomization; two arms have a multiple crossover design (with different intervention orders to the crossover) and one arm has no order prescribed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Trial ABCCBA (Experimental): Participants in Arm 1 will receive a Personalized Trial of the 3 stress management interventions in an ABCCBA treatment order, where A=mindfulness meditation, B=yoga, and C=brisk walking. Participants in this arm will be prompted to complete 30-minute stress management sessions during applicable treatment weeks. A link to the stress management video will be delivered via text 3 times per week to the participant during applicable intervention periods in the personalized trial arms. Participants will be limited to three views of study-provided stress management content each week.
  Interventions: Behavioral: Personalized Trial ABCCBA
- Personalized Trial CBAABC (Experimental): Participants in Arm 2 will receive a Personalized Trial of the 3 stress management interventions in a CBAABC treatment order, where A=mindfulness meditation, B=yoga, and C=brisk walking. Participants in this arm will be prompted to complete 30-minute stress management sessions during applicable treatment weeks. A link to the stress management video will be delivered via text 3 times per week to the participant during applicable intervention periods in the personalized trial arms. Participants will be limited to three views of the study-provided stress management content each week.
  Interventions: Behavioral: Personalized Trial CBAABC
- Standard Care (Active Comparator): Participants in Arm 3 will receive Standard Care of the 3 stress management techniques (mindfulness meditation, yoga, and brisk walking). Participants will receive access to the same number of views of the mindfulness meditation, yoga, and brisk walking content given to participants randomized in Arm 1 and Arm 2. However, they will not be prompted to complete any session according to a randomization sequence. A link to the stress management video will be delivered via text 1 time per week to the participant. Participants will be limited to 36 total views of study-provided stress management content (12 total views per stress management technique).
  Interventions: Behavioral: Stress Management Techniques with No Randomization Sequence (or order)

INTERVENTIONS:
Behavioral: Personalized Trial ABCCBA — Participants will receive links for 30-minute videos for all three interventions, for 2 weeks each, 3 times per week, in a specified order (ABCCBA), where A=mindfulness meditation, B=yoga, and C=brisk walking.
  Arms: Personalized Trial ABCCBA
Behavioral: Personalized Trial CBAABC — Participants will receive links for 30-minute videos for all three interventions, for 2 weeks each, 3 times per week, in a specified order (CBAABC), where A=mindfulness meditation, B=yoga, and C=brisk walking.
  Arms: Personalized Trial CBAABC
Behavioral: Stress Management Techniques with No Randomization Sequence (or order) — Participants will have access to all 30-minute videos for A=mindfulness meditation, B=yoga, and C=brisk walking, during the 12-week phase of the study. They will be limited to 12 total views per stress management technique.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to determine if an N-of-1 study design, or within-subject trials that the investigators are calling "Personalized Trials" can improve health outcomes over standard practice for common stress management techniques. This study uses three different stress management interventions to improve individual self-report of perceived stress: guided mindfulness meditation, guided yoga, and guided brisk walking. Arm 1 (n=53) and Arm 2 (n=53) of the trial will deliver the interventions using a Personalized Trial (within-subject, single N, cross-over trial) format. Participants in Arm 3 of the trial (N=106) will be offered the same number of interventions but will not be required to follow the established N-of-1 Personalized Trials framework. At the end of their Personalized Trial, participants in Arms 1 and 2 will receive a summarized report with personalized feedback. Participants in Arm 3 will also receive a report, but with summarized data . Both arms will receive 2 additional weeks of the stress management intervention of their choosing, while continuing to answer daily assessments and wear a Fitbit device. At the end of the study, a final survey will be sent assessing satisfaction with the study.

DETAILED DESCRIPTION:
The purpose of this study is to determine if an N-of-1 (within-subject, single N, cross-over trial) study design, or what the investigators are calling "Personalized Trials" can improve health outcomes over standard practice for common stress management techniques, and can have widespread use in future research and clinical practice to address high public health burdens with a high heterogeneity of treatment response. This study is informed by three previously conducted feasibility pilots of methods to remotely implement Personalized Trials. This current study uses three different stress management interventions to improve individual self-report of perceived stress: guided mindfulness meditation, guided yoga, and guided brisk walking. Participants randomized to Arm 1 (N=53) and Arm 2 (N=53) will receive Personalized Trials stress management interventions (with arms receiving different order of interventions), whereas participants randomized to Arm 3 (N=106) will receive interventions but will not be required to follow the Personalized Trials format. All participants will begin with a 2-week run-in period, where no stress management interventions are given, but data are collected, including daily surveys and Fitbit-derived sleep and activity data, to obtain a baseline average for later statistical comparison. After successful completion of the baseline period, participants will be randomized to receive either one of two orders of 12-weeks of a Personalized Trial or self-directed (standard care) experience, where they can test 3 different stress management techniques in any order they choose while continuing to answer daily assessments and wearing their Fitbit device. At the end of the 12 weeks, all participants will continue to answer daily surveys and wear their Fitbit device for 2 weeks with no experimenter provided intervention, while the study team creates a report containing the individual's observed data. This report will be sent to each participant in all arms, and participants will have the opportunity to select one stress management technique to continue with for 2 additional weeks. After selection, participants will receive six additional sessions of their chosen treatment and will be observed for engagement in these additional wellness sessions. Participants will also be asked to complete daily survey assessments and Fitbit wear for these two additional weeks. At the end of the 18-week study, a final survey will be sent assessing satisfaction with the study. A random sample of 10% of participants from each arm will be asked to participate in a qualitative interview to discuss their experiences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* English speaking
* Self-report of perceived stress raw score of 20 or higher using the Perceived Stress Scale (PSS)
* Owns and can regularly access a smartphone capable of receiving text messages and accessing the internet
* Can regularly wear a Fitbit device
* Lives in the United States

Exclusion Criteria:

* Age < 18 years old
* Women who are pregnant
* Does not speak English
* Does not own or cannot regularly access a smartphone capable of receiving text messages
* Cannot regularly wear a Fitbit device
* Deemed unable to complete the study protocol as a result of cognitive impairment, severe medical or mental illness, or active or prior substance abuse
* Planned surgeries 6 months from study start date
* Individuals who have been previously told by a doctor to not engage in brisk walking 30 minutes, three times per week
* Individuals who have been previously told by a doctor to not engage in yoga
* Lives outside the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Between-Arm Difference in Change in Ecological Momentary Assessment (EMA) of Stress. | : EMA stress will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) during follow-up period (13-18 weeks).
  Stress will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their stress on a scale of 0 (low) to 10 (high). Levels of EMA stress will be aggregated within the baseline assessment period and during the follow-up period to generate an overall mean and standard deviation for each period. The change in EMA stress between baseline and follow-up will be calculated by subtracting these aggregated means. The difference in change in EMA stress between baseline and follow-up periods will be compared between the personalized arms (Arm 1 and 2) and the standard of care arm (Arm 3) using a two-sample t-test and Generalized Linear Mixed Model analyses.

SECONDARY OUTCOMES:
Change in Mean Within-Subject Difference in Weekly Perceived Stress. | Perceived stress will be assessed weekly during the baseline assessment period (2 weeks) during follow-up period (13-18 weeks).
  Weekly perceived stress will be assessed with the 10-item Perceived Stress Scale (PSS-10), modified to be delivered to assess the prior week rather than the prior month. The minimum total score possible is 0 and the maximum total score possible is 40. Higher values represent higher level of stress. Levels of weekly perceived stress will be aggregated within the baseline assessment period and during the follow-up period to generate an overall mean and standard deviation for each period. The change in weekly perceived stress between baseline and follow-up will be examined using Generalized Linear Mixed Model analyses.
Agreement of Intervention Selection Between Participant and Researcher. | Assessed after completion of follow-up (18 weeks from baseline).
  At the end of the intervention in the personalized trial arms (Arm 1 & Arm 2), personalized trial data will be used to identify which intervention (mindfulness, yoga, or walking) was most effective at reducing stress. This recommendation will be presented in a personalized report sent after completion of the intervention. The number of participants in the personalized trial arms who select this recommended intervention during follow-up relative to the total number of participants in Arms 1 & 2 will be presented as a proportion, with a higher proportion indicating greater levels of agreement.
Mean System Usability Score (SUS). | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  The SUS is a validated 10-item questionnaire that asks users to score each item on a Likert scale from Strongly Disagree (rating of 1) to Strongly Agree (rating of 5). The SUS will be presented to the participant as addressing the ease of use, complexity, consistency of the Personalized Trials system as a whole, from recruitment to receipt of the report. Individual results are calculated to arrive at a composite measure out of 100. Participant SUS scores will be averaged together and an overall mean will be reported with standard deviation. Higher scored values correlate to a more usable system, and therefore a better outcome.
Participant Satisfaction with Personalized Trial Components. | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  Participants will rate their satisfaction with the Trial overall and with individual elements of the trial in a satisfaction survey. Satisfaction items are not part of an already existing scale but were developed to assess participant satisfaction with specific elements of the current study and the trial overall. Participants will rate their satisfaction on a scale of 1 to 5, with higher numbers indicating greater levels of satisfaction. Means and standard deviations will be reported for each element of satisfaction.
Within-Subject Difference in Ecological Momentary Assessment (EMA) of Stress. | EMA fatigue will be assessed 3 times daily via text message during the baseline assessment period (2 weeks), during intervention period (12 weeks) and during follow-up period (4 weeks), 18 weeks total.
  Stress will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their stress on a scale of 0 (low) to 10 (high). Levels of EMA stress will be aggregated within the baseline assessment period, in each of the treatment periods (yoga, meditation, guided walking), and during the follow-up period to generate an overall mean and standard deviation for each period. Changes in EMA stress over the course of the entire study will be evaluated using Generalized Linear Mixed Model analyses.
Within-Subject Difference in Ecological Momentary Assessment (EMA) of Fatigue. | EMA fatigue will be assessed 3 times daily via text message during the baseline assessment period (2 weeks), during intervention period (12 weeks) and during follow-up period (4 weeks), 18 weeks total.
  Fatigue will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their fatigue on a scale of 0 (low) to 10 (high). Levels of EMA fatigue will be aggregated within the baseline assessment period and in each of the treatment periods (yoga, meditation, guided walking) to generate an overall mean and standard deviation for each period. Changes in EMA fatigue over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Within-Subject Difference in Ecological Momentary Assessment (EMA) of Pain. | EMA pain will be assessed 3 times daily via text message during the baseline assessment period (2 weeks), during intervention period (12 weeks) and during follow-up period (4 weeks), 18 weeks total.
  Pain will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their pain on a scale of 0 (low) to 10 (high). Levels of EMA pain will be aggregated within the baseline assessment period and in each of the treatment periods (yoga, meditation, guided walking) to generate an overall mean and standard deviation for each period. Changes in EMA pain over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Within-Subject Difference in Ecological Momentary Assessment (EMA) of Mood. | EMA mood will be assessed 3 times daily via text message during the baseline assessment period (2 weeks), during intervention period (12 weeks) and during follow-up period (4 weeks), 18 weeks total.
  Mood will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their mood on a scale of 0 (poor) to 10 (excellent). Levels of EMA mood will be aggregated within the baseline assessment period and in each of the treatment periods (yoga, meditation, guided walking) to generate an overall mean and standard deviation for each period. Changes in EMA mood over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Within-Subject Difference in Ecological Momentary Assessment (EMA) of Concentration. | EMA concentration will be assessed 3 times daily via text message during the baseline assessment period (2 weeks), during intervention period (12 weeks) and during follow-up period (4 weeks), 18 weeks total.
  Concentration will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their concentration on a scale of 0 (low) to 10 (high). Levels of EMA concentration will be aggregated within the baseline assessment period and in each of the treatment periods (yoga, meditation, guided walking) to generate an overall mean and standard deviation for each period. Changes in EMA concentration over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.
Within-Subject Difference in Ecological Momentary Assessment (EMA) of Confidence. | EMA fatigue will be assessed 3 times daily via text message during the baseline assessment period (2 weeks), during intervention period (12 weeks) and during follow-up period (4 weeks), 18 weeks total.
  Confidence will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their confidence on a scale of 0 (low) to 10 (high). Levels of EMA confidence will be aggregated within the baseline assessment period and in each of the treatment periods (yoga, meditation, guided walking) to generate an overall mean and standard deviation for each period. Changes in EMA confidence over the course of the study will be evaluated using Generalized Linear Mixed Model analyses.

OTHER OUTCOMES:
Within-Subject Difference in Fitbit Device-Recorded Daily Steps. | Daily steps will be assessed consistently via Fitbit device during the baseline assessment period (2 weeks), during intervention period (12 weeks) and during follow-up period (4 weeks), 18 weeks total.
  Daily step counts will be assessed by a Fitbit device. Daily step counts will be aggregated within the baseline assessment period and in each of the treatment periods (yoga, meditation, guided walking) to generate an overall mean and standard deviation for each period. Mean daily steps will be compared to baseline using three paired-samples t-tests (yoga vs baseline, meditation vs baseline, guided walking vs baseline). Daily steps values over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Within-Subject Difference in Fitbit Device-Recorded Nightly Sleep. | Nightly sleep duration will be assessed consistently via Fitbit device during the baseline assessment period (2 weeks), during intervention period (12 weeks) and during follow-up period (4 weeks), 18 weeks total.
  Nightly sleep duration will be assessed by a Fitbit device. Sleep duration will be aggregated within the baseline assessment period and in each of the treatment periods (yoga, meditation, guided walking) to generate an overall mean and standard deviation for each period. Mean sleep duration will be compared to baseline using three paired-samples t-tests (yoga vs baseline, meditation vs baseline, guided walking vs baseline). Sleep duration values over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Mean Participant Survey Adherence Rate. | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  For each participant of the proportion of surveys measures completed (both daily and weekly surveys) will be calculated. Completion rates across all participants will be reported with means and standard deviations.
Mean Participant Ecological Momentary Assessment (EMA) adherence rate. | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  For each participant of the proportion of EMA measures completed will be calculated. Completion rates across all participants will be reported with means and standard deviations.
Mean Fitbit Device Adherence Rate. | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  For each participant, the proportion of days where the Fitbit device was worn will be calculated. Completion rates across all participants will be reported with means and standard deviations.
Mean Participant Fitbit Sleep Rate. | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  For each participant, the average days of participant-observed sleep data, defined as recorded sleep and wake cycles, will be calculated across all participants with means and standard deviations.
Mean Participant Personalized Trial Intervention Adherence Rate. | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  For each participant, the intervention adherence rate, defined as unique video views of the appropriate recorded intervention during the assigned interventions, will be calculated and reported across all applicable individuals with means and standard deviations.
Mean Participant Standard Care Intervention Adherence Rate. | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  For each participant, the intervention adherence rate, defined as unique video views of the appropriate recorded intervention during the assigned interventions, will be calculated and reported across all applicable individuals with means and standard deviations.
Mean Participant Selection Adherence Rate. | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  For each participant, the follow-up period adherence rate, defined as unique video views of the appropriate recorded intervention during the assigned follow-up period, will be calculated and reported across all individuals with means and standard deviations.
Descriptive Content of Qualitative Interview Data | Assessed once after the results report has been sent to the participant after completion of the trial (18 weeks from baseline).
  After completion of the trial, a random sample of 10% of participants from each arm will be asked to participate in 60-minute qualitative interviews to discuss their experiences. Descriptive content from these recorded and transcribed interviews will be analyzed and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, PhD, MASc, Principal Investigator — Northwell Health
Locations (1):
- Institute of Health System Science, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary.
  Supporting Information: Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
  Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Goodwin AM, Miller D, D'Angelo S, Perrin A, Wiener R, Greene B, Romain AN, Arader L, Chandereng T, Kuen Cheung Y, Davidson KW, Butler M. Protocol for randomized personalized trial for stress management compared to standard of care. Front Psychol. 2023 Sep 19;14:1233884. doi: 10.3389/fpsyg.2023.1233884. eCollection 2023. PMID 37794909

DOCUMENTS (1):
  • Informed Consent Form (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT05408832/ICF_000.pdf